CLINICAL TRIAL: NCT03665857
Title: A School-based Multicomponent Intervention Study for Preventing Excessive Weight Gain Among Primary School Students
Brief Title: Childhood Obesity Intervention Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Hai-Jun Wang, Professor in Department of Maternal and Child Health, School of Public Health, Peking University, Peking University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2016YFC1300204
Record Dates: First submitted 2018-09-03; First posted 2018-09-11 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Pediatric Obesity
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessors measuring childrens' weight and height will be blinded at follow-up phases.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- multicomponent intervention (Experimental): Schools in the intervention arm will receive a multicomponent intervention at the school-, parent- and student-level, with a mobile application to promote the collaboration between investigators, school teachers, parents and students.
  The school-level intervention elements will include school policies and health education for teachers.
  The parent-level intervention elements will include health education for parents and promoting students' physical activity at home.
  The student-level intervention elements will include health education for students, promoting students' physical activity in school and monthly monitoring of weight and height.
  Interventions: Behavioral: a multicomponent intervention
- usual-care control (No Intervention): Schools assigned to the control group will have usual education provision throughout their participation in the trial, and after finishing the study they will be offered the health education package, policy suggestion and materials as the schools in the multicomponent intervention group.

INTERVENTIONS:
Behavioral: a multicomponent intervention — 1. School-level policies Students will not be allowed to drink sugar-sweetened beverage or eat unhealthy snacks in schools and drinking water will be advocated.
  2. Monitoring of students' weight and height Students will be monitored their weight and height monthly.
  3. Promotion of physical activity Students will be required to perform at least 60 minutes of moderate to vigorous physical activity each day in school and increase their physical activity outside school (reaching 30 minutes per weekday and one hour per weekend day).
  4. Health education activities Health education activities will be provided for students (10 sessions, 40 minutes per session, 2-3 weeks once), parents and school teachers.
  5. The mobile application The mobile application will disseminate health education knowledge among students, parents and teachers, monitor and provide feedback of students' BMI status and diet and physical activity behaviors.
  Arms: multicomponent intervention

SUMMARY:
Globally, childhood overweight and obesity is a public health problem. Although the rising trend in children's body mass index (BMI) has plateaued in some high-income countries, it has accelerated in low- and middle-income countries. It is especially true amongst Chinese children with the annual increase rate of obesity during 2010-2014 greater than any other periods from 1985 to 2010.

With the dramatic economic development in China, children are now growing up in an increasingly 'obesogenic' environment. For example, the availability and ubiquity of computers and smart phones promote sedentary time, and access to energy dense food and sugar sweetened beverages is now widespread. Effective childhood obesity intervention is urgently needed in China. Although over 20 intervention studies for overweight/obesity among children and adolescents have been conducted in China since the 1990s, most of them had moderate or serious methodological weaknesses. For example, they did not report the number of students, schools or districts initially approached to participate, raising the possibility of selection and recruitment bias. Additionally, although they stated the allocation of intervention and control were randomized, no description of the method of randomization was reported.

Given the relative lack of high-quality interventions for childhood overweight/obesity, the investigators designed a cluster randomized controlled trial to assess the effectiveness of a multicomponent one-academic-year intervention among 24 primary schools (approximately 1200 students) in the eastern (Beijing), middle (Shanxi) and western (Xinjiang) part of China.

The study aims to identify: 1) whether the school-based intervention will be effective for preventing excessive weight gain among children; 2) whether the intervention will be beneficial for improving healthy eating, physical activity and reducing sedentary behaviors among children.

ELIGIBILITY:
1. Eligibility criteria for schools The trial recruited a total of 24 schools. A convenience sample of 8 schools were selected from Beijing, Shanxi (Changzhi City) and Xinjiang (Urumqi City) respectively.

1. Inclusion Criteria for schools:

   * school leader agreeing to implement this intervention; requiring school teachers who can implement this intervention (e.g. school doctors, physical education teachers, physical education teachers, etc.); having at least 50 children from Grade 4 (at the start of the intervention) per school;having a even number of schools within each district.
2. Exclusion Criteria for schools:

   * boarding schools;schools solely for children with special skills; schools of minor ethnic groups; similar programme (focus on weight gain prevention) would be conducted in schools during the study period; schools having a cancelling or relocation plan during the study period.

     2. Eligibility criteria for classes One class per school will be selected if the estimated number of students enrolled in the programme is no less than 40 within the selected class; two classes per school will be selected if the estimated number of students enrolled in the programme is less than 40 within the selected class.

     3. Eligibility criteria for students Eligible children will be those whose primary caregivers will provide written consent to participate the study. After collecting students' medical history from their parents, we will exclude individuals suffering from or having a history of any cardiovascular and metabolic diseases, asthma and disabilities that limit their ability to perform physical activity.

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1392 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2021-04-29 (Actual)

PRIMARY OUTCOMES:
Students' BMI change immediately after the intervention completion | at end of the 8-month intervention
  the difference between arms in the change of students' BMI immediately after the intervention completion

SECONDARY OUTCOMES:
Students' BMI change one year after the intervention completion | at 15 months following the end of the intervention
  the difference between arms in the change of students' BMI one year after the intervention completion
Students' BMI-Z change | 1. at end of the 8-month intervention; 2. at 15 months following the end of the intervention
  use BMI to calculate BMI-Z score based on WHO growth chart
The change of prevalence of childhood overweight/obesity | 1. at end of the 8-month intervention; 2. at 15 months following the end of the intervention
  define childhood overweight or obesity based on international BMI percentile criteria (IOTF)
The change of incidence of childhood overweight/obesity | 1. at end of the 8-month intervention; 2. at 15 months following the end of the intervention
  define childhood overweight or obesity based on international BMI percentile criteria (IOTF)
The change of students' waist circumference | 1. at end of the 8-month intervention; 2. at 15 months following the end of the intervention
  measure waist circumference
The change of students' waist-to-hip circumference ratio | 1. at end of the 8-month intervention; 2. at 15 months following the end of the intervention
  measure waist circumference and hip circumference to calculate waist-to-hip circumference ratio
The change of both systolic and diastolic blood pressures among students | 1. at end of the 8-month intervention; 2. at 15 months following the end of the intervention
  measure systolic and diastolic blood pressure by using electronic sphygmomanometer
The change of body fat percentage among students | at end of the 8-month intervention
  measure body fat percentage by bioelectrical impedance analysis
The change of one-minute rope skipping test outcomes among students | at end of the 8-month intervention
  count the number of one-minute rope skipping
The change of one-minute sit-up test outcomes among students | at end of the 8-month intervention
  count the number of one-minute sit-up test
The change of endurance run (50 metre*8) test outcomes among students | at end of the 8-month intervention
  record the time of endurance run (50 metre*8)
The change of standing long jump test outcomes among students | at end of the 8-month intervention
  measure the distance of standing long jump
The change of students' knowledge related to energy balance | at end of the 8-month intervention
  We will use a self-designed questionnaire including 8 items to assess the change of students' knowledge related to energy balance. For example, we will ask students, "Is it right that drinking sugar-sweetened beverage cannot substitute drinking water." Three choices will be provided (Right; Wrong; Not clear).
The change of students'duration of moderate-to-vigorous physical activity | at end of the 8-month intervention
  Questions were designed based on a validated 7-day physical activity questionnaire. Kappa values for a two-week test-retest ranged from 0.46 to 0.79.
The change of students' eating behavior | at end of the 8-month intervention
  We will use a parent-rated "Children Eating Behavior Questionnaire" (CEBQ) to assess students' eating behaviors, including responsiveness to food, enjoyment of food etc. This 35-item instrument has been shown relatively good reliability.
The change of students' sedentary behavior | at end of the 8-month intervention
  We will use a self-designed questionnaire to ask the average duration of doing homework, watching television and playing electronic devices per day during the last week, respectively.
The change of school-level policies for childhood overweight/obesity | at end of the 8-month intervention
  We will use a self-designed questionnaire to measure school obesity-related policies involving school administration, health education, management of overweight or obesity, communication with the families of students and school lunch.

OTHER OUTCOMES:
The stage of change related to weight reduction behavior | at end of the 8-month intervention
  We will use two items to assess it. First, we will ask "Have you taken action to reduce your weight during the last three months?" Yes/no choices will be provided. And then, we will ask "Do you intend to reduce your weight currently?" This item will be provided 5 choices from "completely not intend" to "intend very much".

CONTACTS AND LOCATIONS:
Overall Officials: Hai-Jun Wang, PhD, Principal Investigator — Peking University
Locations (1):
- Department of Maternal and Child Health, School of Public Health, Peking University, Beijing, China

REFERENCES:
- [Derived] Yan S, Zhou S, Guo X, Lyu J, Wang H, Fang H, Wang HJ. Economic evaluation of a multi-component obesity prevention intervention in Chinese primary schools. BMC Med. 2025 Nov 24;23(1):653. doi: 10.1186/s12916-025-04451-x. PMID 41286848
- [Derived] Liu Z, Gao P, Gao AY, Lin Y, Feng XX, Zhang F, Xu LQ, Niu WY, Fang H, Zhou S, Li WH, Yuan JH, Xu CX, Wu N, Li HJ, Wen LM, Patton GC, Wang HJ, Wu YF. Effectiveness of a Multifaceted Intervention for Prevention of Obesity in Primary School Children in China: A Cluster Randomized Clinical Trial. JAMA Pediatr. 2022 Jan 1;176(1):e214375. doi: 10.1001/jamapediatrics.2021.4375. Epub 2022 Jan 4. PMID 34747972
- [Derived] Liu Z, Wu Y, Niu WY, Feng X, Lin Y, Gao A, Zhang F, Fang H, Gao P, Li HJ, Wang H; study team for the DECIDE-children study. A school-based, multi-faceted health promotion programme to prevent obesity among children: protocol of a cluster-randomised controlled trial (the DECIDE-Children study). BMJ Open. 2019 Nov 2;9(11):e027902. doi: 10.1136/bmjopen-2018-027902. PMID 31678935